CLINICAL TRIAL: NCT01403714
Title: A Randomized Trial of Percutaneous Renal Intervention With Stenting for Patients With Heart Failure and Hemodynamically Significant Renal Artery Stenosis
Brief Title: Study of Percutaneous Renal Artery Intervention for Patient With Heart Failure
Acronym: STRETCH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit eligible subjects
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 813650
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Heart Failure
Keywords: acute heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Management (No Intervention): Patients may be randomized to medical management alone
- Renal Artery Stenting (Active Comparator): Those patients with recent heart failure exacerbations that cannot be attributed to poor left ventricular function and have a hemodynamically significant renal artery stenosis may be randomized to renal artery stenting
  Interventions: Procedure: Renal Artery Stenting

INTERVENTIONS:
Procedure: Renal Artery Stenting — If the patient has a hemodynamically significant renal artery stenosis, and they are randomized to renal artery stenting, they will undergo renal artery stenting
  Arms: Renal Artery Stenting

SUMMARY:
This study will address the role of percutaneous renal intervention for a hemodynamically significant renal artery stenosis in patients with heart failure exacerbations. Current guidelines suggest evaluation for renal artery stenosis in patients with pulmonary edema or heart failure that cannot be attributed to poor left ventricular function. While case series have suggested benefit to percutaneous intervention in patients with heart failure, no randomized study has addressed the potential benefit of renal stenting for heart failure patients. Two large randomized trial of renal stenting for hypertension or poor kidney function failed to show benefit in patients with intermediate renal artery lesions. No evaluation of the potential hemodynamic significance of the lesions was performed prior to randomization. The investigators will enroll patients with heart failure exacerbations not attributable to declining left ventricular function, valvular disease, acute coronary syndrome, or heart transplant rejection, who on non-invasive imaging appear to have renal artery stenosis. After routine invasive assessment, including renal angiography and pressure-wire assessment, patients with hemodynamically significant renal artery stenoses will be randomized to stent implantation or medical therapy. Patients will then be followed to determine whether stenting impacts cardiac mortality or hospitalization for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 or older referred for invasive evaluation of possible renal artery stenosis will be screened for enrollment.

Patients must be inpatients admitted for heart failure exacerbation, or have been admitted to a hospital for heart failure exacerbation within the past 90 days. Heart failure is defined as physician documentation or report of any of the following clinical symptoms of heart failure described as dyspnea on exertion, dyspnea occurring in the supine position, fluid retention; or the description of rales, jugular venous distension, pulmonary edema on physical exam, or pulmonary edema on chest x-ray; without being clearly attributable to liver, kidney, or lung disease. Patients must have one of the following: 1. an ejection fraction of 50%; 2. an ejection fraction of 25-50% in the setting of a systolic blood pressure of at least 160 mmHg; or 3. an ejection fraction of 25-50% and a systolic blood pressure of at least 140 mmHg while being treated with at least 2 antihypertensive medications. Patients who meet these criteria and have a proven hemodynamically significant renal artery stenosis (as described in the procedure section) will be included

Exclusion Criteria:

Patients with heart failure from structural heart disease (including greater than moderate dysfunction of the mitral or aortic valve), acute coronary syndrome, post-partum cardiomyopathy, or acute rejection of a transplanted heart will be excluded. Patients who are considered unlikely to survive to hospital discharge will be excluded. Patients with fibromuscular dysplasia, prior renal stenting, or anatomy unsuitable for renal stenting (i.e. prior vascular surgery making stent delivery impossible) will be excluded. Patients who are unable to take aspirin and clopidogrel will be excluded. Patients with a creatinine clearance <30 mL/min or a history of renal transplantation will be excluded. Pregnant women will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
heart failure | one year
  The primary outcome will be the incidence of cardiac mortality or readmission for heart failure after one year.

SECONDARY OUTCOMES:
hospitalizations | five years
  Secondary analyses will include all-cause mortality, all hospitalizations, changes in echocardiographic parameters, changes in heart failure class, changes in renal function, and changes in blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wilensky, M.D., Principal Investigator — University of Pennsylvania; Zachary Gertz, M.D, Study Director — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States